CLINICAL TRIAL: NCT02631954
Title: Phase I Clinical Trial for Comparison of Pharmacokinetic Characteristics of Vorico Injection 200mg(Voriconazole) and Vfend® IV 200mg for Single Dose Crossover Intravenous Infusion in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 151HPS14014
Record Dates: First submitted 2015-12-13; First posted 2015-12-16 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2016-01

CONDITIONS: Aspergillus Infections; Candida Infections; Fungal Infections
MeSH Terms: conditions — Aspergillosis; Candidiasis; Mycoses | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TR Group (Experimental): Test drug: Vorico Injection 200mg(Voriconazole) Wash out: 7 days Reference drug: Vfend® IV 200mg
  Interventions: Drug: Vorico Injection 200mg(Voriconazole); Drug: Vfend®(Voriconazole) IV 200mg
- RT group (Experimental): Reference drug: Vfend® IV 200mg Wash out: 7 days Test drug: Vorico Injection 200mg(Voriconazole)
  Interventions: Drug: Vorico Injection 200mg(Voriconazole); Drug: Vfend®(Voriconazole) IV 200mg

INTERVENTIONS:
Drug: Vorico Injection 200mg(Voriconazole) — Vorico Injection 200mg(Voriconazole) to administered intravenously once
Drug: Vfend®(Voriconazole) IV 200mg — Vfend®(Voriconazole) IV 200mg to administered intravenously once

SUMMARY:
Phase I Clinical Trial for Comparison of Pharmacokinetic Characteristics of Vorico Injection 200mg(Voriconazole) and Vfend® IV 200mg for Single Dose Crossover Intravenous Infusion in Healthy Volunteers

DETAILED DESCRIPTION:
To healthy volunteers subjects of twenty four(24), following treatments are administered dosing in each period injected wash-out period is a minimum of 7days. Treatment A(Test Drug): Vorico Injection 200mg(Voriconazole) for Single Dose Treatment B(Reference Drug): Vfend® IV 200mg for Single Dose Pharmacokinetic blood samples are collected up to 24hrs.

Safety and pharmacokinetic are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy person whose age is in between 19 to 55 during the screening tests
2. Whose weight is more than 55 kg, BMI is over 18.5 and under 30.0 during the screening test. (BMI (kg/m2) = weight (kg) / {height (m)}2)
3. Who is completely informed and understand about this clinical trial, voluntarily participating it, and signed to follow the given instructions
4. Who is proven to fit into the clinical trial following by physical examination, ECG (electrocardiogram), clinical laboratory test, medical examination
5. Who agreed to do birth control during testing

   * A male who did not have vasectomy has to follow the clinically proven contraceptive methods* listed under, and who agreed not to donate sperm during the test

     * Clinically proven contraceptive method: intrauterine device (ex. Lippes Loop, Minera), chemical contraceptive (spermicides) for use with physical contraceptive method (males or females), contraceptive implants (ex. Implanon), tubal ligation or laparoscopy (common methods of tubal ligation)
   * A woman of childbearing age who agreed on constant use of a medically disproven Dual Protection method** and spermicides except hormonal contraceptive, and who also agreed not to breastfeed.

     * A Dual Protection method: use of condoms, the Intrauterine Contraceptive Device, the diaphragm, the cervical cap, in the case where a sexual partner had vasectomy over 3 months ago (from the date of initial screening) or a sexual partner had been medically diagnosed sterile.

Exclusion Criteria:

1. A person who has a history of clinically significant cardiovascular, respiratory, liver, kidney, endocrine system, immune system, urinary system diseases, blood-tumor diseases, mental illness.
2. Who has a history of hypersensitivity reactions to antifungal drugs including voriconazole or similar series or other excipient ingredients (aspirin, antibiotics, etc.)
3. Who has genetics issues on galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption
4. Who has a history of gastrointestinal disease (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (other than simple appendectomy and herniotomy)
5. A person whose electrocardiogram value includes QTc > 440 msec, PR < 110 msec or PR > 200 msec, QRS < 60 msec or QRS > 110 msec after screening, or who show clinically significant opinion.
6. Who falls under the following results

   1. AST, ALT are exceeded over 1.5x the upper limit of the normal range
   2. Total bilirubin is exceeded over 1.5x the upper limit of the normal range
7. Who shows the vital sign values of more than 140 mmHg or less than 90 mmHg in systolic pressure or more than 100 mmHg or less than 60 mmHg in diastolic blood pressure
8. Who has history of drug abuses or shows a positive result in the urinary drug screen
9. Who took any prescribed drugs, medicinal plants within the 2 weeks before the first day of dosing or takes any over-the-counter drugs or vitamin supplements within 1 week (but, if other conditions are met, they can still participate in the clinical test through the researcher's judgment)
10. Who took other investigational drugs or bioequivalence drugs within 3 months before the first day of dosing
11. Who participated in whole blood donation within 2 months before the first of dosing, or platelet donations within 1 months. Who received blood a month before the first day of dosing
12. Who constantly drinks alcohol (over 21 units/week, 1 unit = 10 g of pure alcohol) or cannot stop drinking alcohol during the clinical test.
13. Who smokes more than 10 cigarettes per day, or who cannot quit smoking when hospitalized
14. Who absorb caffeinated drinks (coffee, tea (black or green tea), soda, coffee flavored milk, energy drinks, etc.) or cannot stop absorbing them 24 hours before hospitalization until discharging
15. Who takes drug metabolism drug like barbital drugs which inhibit or activate the metabolism or drugs, or who takes one of the following drugs: St. John's Wort, rifabutin, rifampicin, carbamazepine, phenobarbital, high-dose of ritonavir, terfenadine, astemizole, cisapride, pimozide, quinidine, sirolimus, ergot, alkaloid (ergotamine, dihydroergotamine), efavirenz
16. Who was having foods (especially grapefruit or products contain grapefruit) that can influence the drug absorption, distribution, metabolism, and excretion within 7 days from the first day of dosage
17. A woman who is pregnant, shows positive result in serum/urine test, or who is breastfeeding

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

REFERENCES:
- [Derived] Cho SH, Kim CW, Nam MS. Pharmacokinetics and Safety of Two Voriconazole Formulations after Intravenous Infusion in Healthy Korean Volunteers. Infect Chemother. 2020 Jun;52(2):204-211. doi: 10.3947/ic.2020.52.2.204. Epub 2020 May 29. PMID 32468741

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who passed the screening were randomized using IWRS before conducting the clinical trail.
Period: Overall Study
Arm/Group | TR Group | RT Group
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 24 subejcts were used for baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | TR Group | RT Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants] — Population: healthy subjects aged 19 to 55 yesars were selected.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 12 | 12 | 24
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Voriconazole
Description: The blood sampleing coleected from the subjects was analyzed and result was obtained.
Time Frame: 0 , 0.5, 1, 1.25, 1.5, 1.58, 1.67, 1.83, 2, 2.5, 3, 4, 6, 8, 12, 24 hrs
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Reference: Reference: Vfend® IV 200mg drug
  * RT group: Vfend®(Voriconazole) IV 200mg to administered intravenously once at Period I
  * TR group: Vfend®(Voriconazole) IV 200mg to administered intravenously once at Period II
- Test: Test: Vorico Injection 200mg(Voriconazole) drug
  * RT group: Vorico Injection 200mg(Voriconazole) to administered intravenously once at Period II
  * TR group: Vorico Injection 200mg(Voriconazole) to administered intravenously once at Period I
Arm/Group | Reference | Test
Number analyzed (Participants) | 23 | 23
ng/mL | 2433.7 (2456.9) | 1997.0 (406.2)

2. Primary Outcome: AUCt of Voriconazole
Description: The blood sampleing coleected from the subjects was analyzed and result was obtained.
Time Frame: 0 , 0.5, 1, 1.25, 1.5, 1.58, 1.67, 1.83, 2, 2.5, 3, 4, 6, 8, 12, 24 hrs
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Reference | Test
Number analyzed (Participants) | 23 | 23
hr*ng/mL | 6966.17 (2856.10) | 7469.78 (3125.73)

3. Secondary Outcome: Tmax of Voriconazole
Description: The blood sampleing coleected from the subjects was analyzed and result was obtained.
Time Frame: 0 , 0.5, 1, 1.25, 1.5, 1.58, 1.67, 1.83, 2, 2.5, 3, 4, 6, 8, 12, 24 hrs
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Reference | Test
Number analyzed (Participants) | 23 | 23
hr | 1.57 (0.03) | 1.58 (0.04)

4. Secondary Outcome: AUCinf of Voriconazole
Description: The blood sampleing coleected from the subjects was analyzed and result was obtained.
Time Frame: 0 , 0.5, 1, 1.25, 1.5, 1.58, 1.67, 1.83, 2, 2.5, 3, 4, 6, 8, 12, 24 hrs
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Reference | Test
Number analyzed (Participants) | 23 | 23
hr*ng/mL | 8159.24 (4905.05) | 8631.50 (4401.54)

5. Secondary Outcome: AUCt/AUCinf
Description: The blood sampleing coleected from the subjects was analyzed and result was obtained.
Time Frame: 0 , 0.5, 1, 1.25, 1.5, 1.58, 1.67, 1.83, 2, 2.5, 3, 4, 6, 8, 12, 24 hrs
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Reference | Test
Number analyzed (Participants) | 23 | 23
Ratio | 0.94 (0.10) | 0.90 (0.09)

6. Secondary Outcome: Kel (Elemination Rate Constant)
Description: The blood sampleing coleected from the subjects was analyzed and result was obtained.
Time Frame: 0 , 0.5, 1, 1.25, 1.5, 1.58, 1.67, 1.83, 2, 2.5, 3, 4, 6, 8, 12, 24 hrs
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Reference | Test
Number analyzed (Participants) | 23 | 23
1/hr | 0.10 (0.03) | 0.10 (0.04)

7. Secondary Outcome: t1/2
Description: The blood sampleing coleected from the subjects was analyzed and result was obtained.
Time Frame: 0 , 0.5, 1, 1.25, 1.5, 1.58, 1.67, 1.83, 2, 2.5, 3, 4, 6, 8, 12, 24 hrs
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Reference | Test
Number analyzed (Participants) | 23 | 23
hr | 8.42 (4.61) | 7.98 (2.92)

ADVERSE EVENTS:
Time Frame: 1 months
Description: There was no serious AE. A total of 58 AEs out of 24 subjects who took IP more than at least one time, were observed.
  All of the AEs were mild and recovered.
Arm/Group | Reference | Test
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 21/23 | 22/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reference (N=23) | Test (N=24)
photophobia (Eye disorders) | 18 | 21
colour blindness acquired (Eye disorders) | 1 | 0
vision blurred (Eye disorders) | 2 | 0
visual impariment (Eye disorders) | 1 | 1
headache (Nervous system disorders) | 0 | 2
blood glucose increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
urine oxalate increased (Investigations) | 0 | 1
white blood cells urine positive (Investigations) | 1 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
dizziness (Vascular disorders) | 3 | 3
epistaxis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No